CLINICAL TRIAL: NCT05483439
Title: Clinical Study Comparing the Efficacy and Safety of Traditional Herbal Medicine for Cancer Immunotherapy Combined With Neoadjuvant Therapy Versus Neoadjuvant Therapy in Patients With Stage II-III Breast Cancer.
Brief Title: A Study of Immunotherapy Combined With Neoadjuvant Therapy Versus Neoadjuvant Therapy for Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, professor, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shengjing-LCG012
Record Dates: First submitted 2022-07-21; First posted 2022-08-02 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Stage II-III Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cytotoxins; Docetaxel; Epirubicin; Cyclophosphamide; Carboplatin; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunotherapy and neoadjuvant therapy (Experimental): Traditional herbal medicine twice daily combined with neoadjuvant therapy recommended by the guidelines every 3 weeks, for 6 or 8 cycles.
  Interventions: Drug: cytotoxic chemotherapy (docetaxel or epirubicin or cyclophosphamide or carboplatin); Drug: anti-Her2 monoclonal antibody (Trastuzumab, Pertuzumab); Drug: traditional herbal medicine
- neoadjuvant therapy (Other): Only received neoadjuvant therapy recommended by the guidelines every 3 weeks, for 6 or 8 cycles.
  Interventions: Drug: cytotoxic chemotherapy (docetaxel or epirubicin or cyclophosphamide or carboplatin); Drug: anti-Her2 monoclonal antibody (Trastuzumab, Pertuzumab)

INTERVENTIONS:
Drug: cytotoxic chemotherapy (docetaxel or epirubicin or cyclophosphamide or carboplatin) — Drug: cytotoxic chemotherapy (docetaxel or epirubicin or cyclophosphamide or carboplatin)
Drug: anti-Her2 monoclonal antibody (Trastuzumab, Pertuzumab) — anti-Her2 monoclonal antibody (Trastuzumab, Pertuzumab)
Drug: traditional herbal medicine — traditional herbal medicine
  Arms: Immunotherapy and neoadjuvant therapy

SUMMARY:
This is a randomized, open label Phase II neoadjuvant study comparing the efficacy and safety of the combination of traditional herbal medicine for cancer immunotherapy and neoadjuvant therapy versus neoadjuvant therapy in patients with breast cancer.

DETAILED DESCRIPTION:
This is a randomized, open label Phase II neoadjuvant study comparing the efficacy and safety of the combination of traditional herbal medicine for cancer immunotherapy and neoadjuvant therapy versus neoadjuvant therapy in patients with breast cancer. Patients will be randomized (1:1) to one of the two treatment arms: arm 1, combination of traditional herbal medicine for cancer immunotherapy and neoadjuvant therapy for 6 or 8 cycles; arm 2, neoadjuvant therapy 6 or 8 cycles. Patients will undergo surgery after neoadjuvant therapy. Efficacy will be assessed every 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥ 18 but ≤ 75 years;
2. Diagnosis of breast cancer meets the following criteria: Stage II-III patients who meet the 8th edition of AJCC Cancer Staging Manual and meet the indications of neoadjuvant therapy;
3. Diagnosis of breast cancer meets the following criteria: Histologically confirmed invasive breast cancer
4. KPS score≥70
5. The functional level of major organs must conform to the following requirements: Neutrophils (ANC) ≥ 1.5×10^9/L (with no use of growth factors within 14 days); Platelet count (PLT) ≥ 100×10^9/L (with no correct treatment within 7 days ); Hemoglobin (Hb) ≥ 90 g/L (with no correct treatment within 7 days ); Total bilirubin (TBIL) ≤ 1.5×upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3×ULN; Urea nitrogen and creatinine ≤ 1.5×ULN and creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula); Cardiac color Doppler ultrasound: left ventricular ejection fraction (LVEF) ≥ 50%; 12-lead electrocardiogram: QT interval ≤ 480 ms;
6. Patients who participate in the trial voluntarily, sign an informed consent, have good compliance and are willing to comply with the follow-up visit.

Exclusion Criteria:

1. Previously received any anti-tumor therapy (chemotherapy, radiotherapy, molecular targeted therapy, endocrine therapy, etc.);
2. Patients who are concurrently receiving other anti-tumor therapy;
3. Bilateral breast cancer, inflammatory breast cancer, or occult breast cancer;
4. Stage IV breast cancer;
5. Intolerant to herbs or poor compliance;
6. With a history of any malignancies other than breast cancer in the past 5 years, excluding cured cervical carcinoma in situ and melanoma skin cancer;
7. Severe heart, liver, kidney and other important organ dysfunction;
8. Inability to swallow, chronic diarrhea and intestinal obstruction, and having many factors that affect drug administration and absorption;
9. Participated in clinical trials of other drugs within 4 weeks before enrollment;
10. Known history of allergy to the drug components of this regimen; History of immunodeficiency, including HIV positive, HCV, live active hepatitis B or other acquired or congenital immune deficiency diseases, or a history of organ transplantation;
11. Have used drugs that affect immune function within 1 year;
12. Once suffered from any heart disease, including: (1) arrhythmia with clinical significance, (2) myocardial infarction; (3) heart failure; (4) investigator's judgment as not suitable for participating in this trial;
13. Pregnant, lactating women, fertile women with positive baseline pregnancy test or in the entire women of reproductive age who were unwilling to use effective contraception during the trial;
14. According to the investigator's judgment, there are comorbidities (including but) that seriously endanger the patient's safety or affect the patient's ability to complete the study not limited to severe hypertension, severe diabetes, active infection, etc., which cannot be controlled by drugs);
15. A clear past history of neurological or psychiatric disorders, including epilepsy or dementia. The investigator considered the patient unsuitable for the study in any other case.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Total pathological complete response rate (tpCR) | One month after surgery
  The disappearance of all invasive tumours in the breast and axillary lymph nodes

SECONDARY OUTCOMES:
Global health status and functioning subscales | One month after surgery
  Health-related quality of life (HRQoL) was measured using the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core-30 (QLQ-C30; version 3).
Cancer-related fatigue scores | One month after surgery
  Piper Fatigue Scale will be used to measure cancer-related fatigue. The scale scores were measured：at baseline, at the end of cycles 2 and 4, and before surgery. Each score represents the degree of fatigue: a score of 0 means none, 1-3 means mild, 4-6 means moderate, 7-10 means severe.
Adverse events (AE) and serious adverse events (SAE) | Period of neoadjuvant therapy (treatment 1-6 months)
  For adverse events (AE) and serious adverse events (SAE), refer to NCI-CTC AE 5.0 standard.
Disease free survival (DFS) | 5 years
  Disease-free survival (DFS) is the time from the day of enrollment to the first occurrence of recurrent disease, including second primary malignancies in the non-breast area and breast ductal carcinoma in situ.
Five-year overall survival (OS) | 5 years
  Five-year overall survival (OS) is the time from the random date to death due to any cause.
Expression of immune cells | One month after surgery
  Expression of immune cells (T cell, B cell, NK cell )
Expression of cytokines (IL, INF-r, TNF-a) | One month after surgery
  Expression of cytokines (IL, INF-r, TNF-a)

CONTACTS AND LOCATIONS:
Overall Officials: Caigang Liu, doctor, Principal Investigator — Shengjing Hospital
Locations (2):
- China (2):
  - ShengJing ospital of China Medical University, Shenyang, Liaoning
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning